CLINICAL TRIAL: NCT05944497
Title: Changes in Pulse Wave Transit Time and Its Variability Measured From the Ipsilateral First Finger After Placement of Interscalene Brachial Plexus Block
Brief Title: Changes in Pulse Wave Transit Time and Its Variability After Placement of Interscalene Brachial Plexus Block
Status: Completed | Type: Observational
Sponsor: JongHae Kim (Other)
Responsible Party: Sponsor-Investigator, JongHae Kim, Professor, Daegu Catholic University Medical Center
Organization: Daegu Catholic University Medical Center (Other)
Other Study IDs: 2023-01
Record Dates: First submitted 2023-06-28; First posted 2023-07-13 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Interscalene Brachial Plexus Block

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ISBPB group: Interscalene brachial plexus block involving the C5 to C8 nerve roots
  Interventions: Procedure: Interscalene brachial plexus block

INTERVENTIONS:
Procedure: Interscalene brachial plexus block — Using a linear ultrasound transducer connected to an ultrasound machine, the compactly arranged brachial plexus is visualized lateral to the pulsating subclavian artery. The transducer is moved cephalad to visualize the 5th to 8th cervical (C5 to C8) nerve roots located between the anterior and middle scalene muscles. Using an in-plane technique, a block needle is inserted close to a nerve root in a lateral-to-medial direction. The needle is moved to place 0.75% ropivacaine around each nerve root. The C8 nerve root is blocked first, and the C5 nerve root is blocked last. After blocking the four cervical nerve roots, ropivacaine is placed in the intermuscular plane between the sternocleidomastoid and scalene muscles to block the supraclavicular nerves. A total of 26 ml of 0.75% ropivacaine is used for the interscalene brachial plexus block (6 ml per nerve root and 2 ml for the supraclavicular nerves).

SUMMARY:
Pulse wave transit time (PWTT) increases due to decreased arterial vascular tone resulting from sympathetic blockade caused by regional anesthesia. Its oscillation (PWTT variability) also contains information on the interaction between autonomic nervous system and the cardiovascular system. The changes in PWTT and its variability have not been investigated in patients receiving interscalene brachial plexus block (ISBPB). It was hypothesized that ISBPB increases PWTT and reduces low frequency power of PWTT variability.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists status of 1
* Scheduled to receive interscalene brachial plexus block for arthroscopic shoulder surgery

Exclusion Criteria:

* Coagulopathy
* Infection of the skin area for interscalene brachial plexus block
* Peripheral neuropathy or neurologic sequelae in the upper limb ipsilateral to the surgery
* Allergy to local anesthetics or a history of allergic shock
* Contralateral vocal cord palsy, hemidiaphragmatic paresis/paralysis or pneumo/hemo thorax
* Arrhythmias
* Cardiac conduction abnormalities
* A history of medication affecting cardiac conduction
* Ischemic heart disease
* Hypertension
* Diabetes mellitus
* Thyroid disfunction
* Other medical conditions affecting autonomic nervous activity

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Tertiary university medical center
Sampling Method: Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2023-07-31 (Actual); Primary Completion 2024-01-07 (Actual); Study Completion 2024-01-07 (Actual)

PRIMARY OUTCOMES:
Natural-log-transformed low frequency power of pulse wave transit time variability | Between 15 and 20 minutes after block needle insertion
  Calculated by integrating the power spectra of pulse wave transit time variability between 0.04 and 0.15 Hz.

SECONDARY OUTCOMES:
Natural-log-transformed low frequency power of pulse wave transit time variability | During 5 minutes before the end of the acclimatization period
  Calculated by integrating the power spectra of pulse wave transit time variability between 0.04 and 0.15 Hz.
Natural-log-transformed low frequency power of pulse wave transit time variability | Between 5 and 10 minutes after block needle insertion
  Calculated by integrating the power spectra of pulse wave transit time variability between 0.04 and 0.15 Hz.
Natural-log-transformed high frequency power of pulse wave transit time variability | During 5 minutes before the end of the acclimatization period
  Calculated by integrating the power spectra of pulse wave transit time variability between 0.15 and 0.4 Hz.
Natural-log-transformed high frequency power of pulse wave transit time variability | Between 5 and 10 minutes after block needle insertion
  Calculated by integrating the power spectra of pulse wave transit time variability between 0.15 and 0.4 Hz.
Natural-log-transformed high frequency power of pulse wave transit time variability | Between 15 and 20 minutes after block needle insertion
  Calculated by integrating the power spectra of pulse wave transit time variability between 0.15 and 0.4 Hz.
Pulse wave transit time | During 5 minutes before the end of the acclimatization period
  Time difference in milliseconds between the R peak of the electrocardiographic waveform and the peak of the 2nd-derivative photoplethysmographic waveform.
Pulse wave transit time | Between 5 and 10 minutes after block needle insertion
  Time difference in milliseconds between the R peak of the electrocardiographic waveform and the peak of the 2nd-derivative photoplethysmographic waveform.
Pulse wave transit time | Between 15 and 20 minutes after block needle insertion
  Time difference in milliseconds between the R peak of the electrocardiographic waveform and the peak of the 2nd-derivative photoplethysmographic waveform.
Sensory blockade | 20 minutes after block needle insertion
  Assessed by grading the coldness with a 3-level scale consisting of 0 (no cold sensation), 1 (reduced cold sensation), and 2 (normal cold sensation) after applying an alcohol swab to the upper limb dermatomal areas innervated by the C5 to T1 nerve roots.
Motor blockade | 20 minutes after block needle insertion
  The muscle contraction power is rated as 0 (complete block), 1 (partial block), and 2 (no block) for shoulder abduction (axillary nerve), elbow flexion (musculocutaneous nerve), forearm supination (radial nerve), forearm pronation (median nerve), wrist extension (radial nerve), wrist flexion (median nerve), finger abduction (ulnar nerve), thumb abduction (radial nerve), thumb adduction (ulnar nerve), and thumb opposition (median nerve).
Bilateral pupil diameters | Within 1 minute after acclimatization
  Measured using a portable automated monocular infrared pupillometer (PLR-3000, NeurOptics Inc., Irvine, CA, the United States) at 30 Hz for 2 seconds.
Bilateral pupil diameters | 20 minutes after block needle insertion
  Measured using a portable automated monocular infrared pupillometer (PLR-3000, NeurOptics Inc., Irvine, CA, the United States) at 30 Hz for 2 seconds.
Incidence of side effects related to interscalene brachial plexus block | 20 minutes after block needle insertion
  Horner's syndrome, subjective dyspnea, and hoarseness

CONTACTS AND LOCATIONS:
Overall Officials: Jonghae Kim, M.D., Principal Investigator — Daegu Catholic University Medical Center
Locations (1):
- Daegu Catholic University Medical Center, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No
IPD will be available from the primary investigator on reasonable request.